CLINICAL TRIAL: NCT00345722
Title: The Long-Term Effect of Viscous Fibers, Soy Protein, and Plant Sterol Foods in Combination on Serum Cholesterol and Other Risk Factors for Cardiovascular Disease
Brief Title: The Effect of Strawberries in a Cholesterol-Lowering Dietary Portfolio
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: California Strawberry Commission (Other); Almond Board of California (Other); Unilever R&D (Industry); Natural Sciences and Engineering Research Council, Canada (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: REB 03-043C; HC-CT#100934
Record Dates: First submitted 2006-06-26; First posted 2006-06-28 (Estimated); Last update posted 2007-05-08 (Estimated); Status verified 2007-05

CONDITIONS: Hyperlipidemia; Cardiovascular Diseases; Hypercholesterolemia
Keywords: Strawberry; Almond; Soy protein; viscous dietary fibre; plant sterols; portfolio diet; blood lipids; compliance; blood pressure
MeSH Terms: conditions — Hyperlipidemias; Cardiovascular Diseases; Hypercholesterolemia; Patient Compliance

INTERVENTIONS:
Procedure: strawberry dietary intervention

SUMMARY:
The purpose of this study is to determine whether addition of strawberries to a dietary portfolio of cholesterol-lowering foods will improve compliance and so increase the effectiveness of the dietary portfolio in lowering cholesterol and improving cardiovascular risk factors.

DETAILED DESCRIPTION:
We have shown in 1-month metabolic studies that the dietary portfolio can lower cholesterol to the same extent as first generation statins (cholesterol-lowering drugs). In the on-going long-term 'real world' study using this dietary portfolio, only one-third of participants were able to achieve similar cholesterol reductions at the end of 1 year. Varying compliance has been identified as the main issue why the other two-thirds could not achieve a similar level of reduction. We believe the addition of strawberries to this diet, by virtue of their beneficial components (fibre and antioxidants)and by replacement of less desirable foods (fatty deserts), may further improve the CHD risk profile of a very effective cholesterol reduction strategy.

Method:

454 g of strawberries per 2000 kcal per day will be provided for a one-month period to approximately 40-50 subjects on a long-term dietary portfolio study, all of whom have been on the diet for at least 6 months to 1 year. The active dietary components consist of viscous vibers (including oat bran), soy products (including soy milk), almonds and plant sterols (sterol enriched margarine). Strawberry recipes will be used to enhance compliance of these components. Subjects will undergo the study in a randomized crossover design where the control will be the dietary portfolio with additional 65 g oatbran bread (without psyllium) replacing the strawberries.

Bloods will be taken at weeks 0, 2 and 4 of each treatment period; and at one month prior to and after the 8-week study while on the long-term dietary portfolio.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men and postmenopausal women currently enrolled in the long-term dietary portfolio study
* Body mass index <32 kg/m2
* constant body weight over last 6 months preceding the onset of the study
* Fasting LDL cholesterol concentration>4.1 mmol/L at diagnosis

Exclusion Criteria:

* women of child-bearing potential
* major cardiovascular event (stroke or myocardial infarction)
* positive molecular diagnosis of familial hypercholesterolemia
* secondary causes of hypercholesterolemia (hypothyroidism, unless treated & on a stable dose of L-thyroxine, renal or liver disease)
* use of cholesterol-lowering medications
* serum triglycerides >4.5 mmmol/L
* blood pressure > 145/90 mmHg
* diabetes and or major disorders such as liver disease, renal failure or cancer
* major surgery <6 months prior to randomization
* alcohol consumption > 2 drinks per day

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2006-06; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Total cholesterol measured at weeks 0, 2, and 4 of each phase
LDL cholesterol measured at weeks 0, 2, and 4 of each phase
C-reactive protein measured at weeks 0, 2 and 4 of each phase
Blood pressure measured at weeks 0, 2 and 4 of each phase

SECONDARY OUTCOMES:
Apolipoprotein A1 and B measured at weeks 0, 2, and 4 of each phase
Lp(a) measured at weeks 0, 2, and 4 of each phase
Oxidative stress measured at weeks 0, 2, and 4 of each phase
Strawberry intake measured at weeks 0, 2, and 4 of each phase
Compliance to portfolio diet components measured at weeks 0, 2 and 4 of each phase
24 hour urinary potassium measured at weeks 0 and 4 of each phase
24 hour urinary calcium measured at weeks 0 and 4 of each phase

CONTACTS AND LOCATIONS:
Overall Officials: David JA Jenkins, MD PhD DSc, Principal Investigator — Department of Nutritional Sciences, Faculty of Medicine, University of Toronto, 150 College St. Rm 340, Toronto, ON M5S 3E2, Canada
Locations (1):
- Clinical Nutrition & Risk Factor Modification Centre, St. Michael's Hospital Health Centre, Toronto, Ontario, Canada